CLINICAL TRIAL: NCT05433337
Title: "PROSPER-FM-EXT": Prospective Study to Evaluate a Digital Regimen for Fibromyalgia Management: An Extension Study
Brief Title: Prospective Study to Evaluate a Digital Regimen for Fibromyalgia Management: An Extension Study
Acronym: PROSPER-FM-EXT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swing Therapeutics, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Swing-005-EXT
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Intervention Model Description: This is a virtual, single-arm, pragmatic, non-significant risk device study. Study participants will continue to have access to Digital Acceptance and Commitment Therapy (ACT) after the original 12-week study (PROSPER-FM, NCT05243511), in addition to their standard care for fibromyalgia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Digital Acceptance and Commitment Therapy (ACT) Arm (Other)
  Interventions: Device: Digital ACT

INTERVENTIONS:
Device: Digital ACT — Study participants will continue to receive Digital Acceptance and Commitment Therapy in addition to their standard care for fibromyalgia

SUMMARY:
This study is designed as a 9-month extension of the original study (PROSPER-FM). The purpose of the extension study is to assess the long-term (up to 1 year) response to a digital therapy in the treatment of fibromyalgia.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant has completed participation in the PROSPER-FM study and was assigned to the Digital ACT Arm
* Participant is willing and able to comply with all protocol-specified requirements

Key Exclusion Criteria:

* Based on the investigator's judgment, any new diagnosis of acute or chronic disease/condition since participant's enrollment in PROSPER-FM study that may impact the outcome of this study
* Severe depression at the final visit of the PROSPER-FM study (measured by BDI-II)
* Increased risk of suicide on the basis of the investigator's judgment or the Columbia-Suicide Severity Rating Scale ("C-SSRS") at the final visit of the PROSPER-FM study

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-03-05 (Actual)

PRIMARY OUTCOMES:
Patient Global Impression of Change (PGIC) | Month 9
  PGIC scores included are: Very much improved, much improved, minimally improved, no change, minimally worse, much worse, very much worse

SECONDARY OUTCOMES:
Revised Fibromyalgia Impact Questionnaire (FIQ-R) total score | Original Study Baseline to Month 9
  FIQ-R total score ranges between 0-100 with a reduction in score indicating reduced fibromyalgia severity.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Keefe, MD, Principal Investigator — Swing Therapeutics
Locations (1):
- Swing Therapeutics, San Francisco, California, United States

REFERENCES:
- See also: Swing Therapeutics Website — https://www.swingtherapeutics.com/